CLINICAL TRIAL: NCT01382706
Title: Single Arm Phase II Study of Docetaxel and Lapatinib in Metastatic Transitional Cell Carcinoma in Bladder as Second Line Treatment
Brief Title: Docetaxel and Lapatinib in Metastatic Transitional Cell Carcinoma in Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial not progressing toward scientific goals
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4B-10-4; NCI-2011-01108 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Bladder Cancer; Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Docetaxel; Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Immunohistochemistry; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and lapatinib ditosylate PO QD on days 1-21. Courses repeat every 21 days until disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: lapatinib ditosylate; Other: immunohistochemistry staining method; Genetic: fluorescence in situ hybridization; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving docetaxel and lapatinib ditosylate together as second-line therapy works in treating patients with stage IV bladder cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel and lapatinib ditosylate together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of 1250 mg of lapatinib (lapatinib ditosylate) given in combination with docetaxel in prolonging progression-free survival of subjects with metastatic, previously treated transitional cell carcinoma (TCC) relative to historical controls.

SECONDARY OBJECTIVES:

I. To assess the efficacy of 1250 mg of Lapatinib given in combination with docetaxel in the objective response rates and overall survival.

II. To study the tolerability and safety of 1250 mg of lapatinib given in combination with docetaxel by assessing the incidence and nature of Grade 3, 4 and serious adverse events (AEs).

TERTIARY OBJECTIVES:

I. To assess the expression status of epidermal growth factor receptor (EGFR) or human epidermal growth factor receptor 2 (HER-2) in tumor tissue and/or circulating tumor cells (CTCs) as potential predictors of response to therapy.

II. To evaluate the number of CTC's present in 7.5mLs of peripheral blood as a predictor for disease progression and response of treatment in bladder cancer in the setting of combination therapy of lapatinib and docetaxel.

III. To evaluate the effect of lapatinib in human at molecular level by targeting the phosphorylation activity of the AKT/extracellular-regulated kinase (ERK) on pathway prior and during the treatment with lapatinib.

OUTLINE: Patients receive docetaxel intravenously (IV) over 1 hour on day 1 and lapatinib ditosylate orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell carcinoma of the urothelium (also called urothelial cancer); mixed histologies are allowed as long as the predominant histology is TCC; in addition, tumor tissue must be available for evaluation for EGFR and HER2/neu status
* Locally recurrent or advanced, non-resectable or stage IV transitional cell carcinoma
* Must have had prior platinum salt-based chemotherapy for TCC; other prior systemic chemotherapeutic or investigational treatment regimens for TCC are allowed; patient may have had up to three lines of chemotherapy for advanced disease; may have had paclitaxel provided their cancer did not progress while on it, and it was part of an adjuvant or neoadjuvant regimen; prior targeted or biological therapy is permitted except for drugs targeting EGFR and/or HER2; specifically, subjects must meet one or more of the following criteria: (a). Progression after treatment with a regimen that includes a platinum salt (e.g. carboplatin or cisplatin) for Stage IV or recurrent disease OR (b). Disease recurrence within two years (from the date of last dose of chemotherapy or surgery until day the informed consent is signed) of neoadjuvant or adjuvant treatment with a regimen that includes a platinum salt
* Measurable or evaluable disease, as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1; if all sites of measurable or evaluable disease have been irradiated, one site must have demonstrated growth after irradiation
* A left ventricular ejection fraction (LVEF) within normal range as measured by echocardiogram or multi-gated acquisition (MUGA) scan
* Adequate contraceptive method for subjects with reproductive potential (females with reproductive potential must have a negative serum pregnancy test within 7 days of study entry)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* A signed written informed consent
* Due to the experimental nature of lapatinib, female subjects must be one year postmenopausal, surgically sterile, or using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation); male subjects must be surgically sterile or using an acceptable method of contraception during their participation in this study

Exclusion Criteria:

* History of treatment of TCC (in any setting - neoadjuvant, adjuvant or for metastatic disease) with docetaxel
* History of treatment with an EGFR or HER2 targeted agent
* Serum bilirubin more than 1.5 x the upper limit of normal (ULN) except in patients with diagnosis of Gilbert's disease
* Creatinine clearance less than 20 mL/minute (calculated by the Cockcroft-Gault formula)
* Potassium, less than institutional normal level despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium below lower limits of normal despite supplementation
* Baseline liver function test including AST or ALT greater than 2.5 x institutional upper limits of normal.
* Absolute neutrophil count (ANC) less than 1500/uL
* Platelets less than 100/uL
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
* An abnormal left ventricular ejection fraction LVEF as measured by echocardiogram or MUGA scan or other suitable technique
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease more than class 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (Common Terminology Criteria for Adverse Events [CTCAE] grade 3) or asymptomatic sustained ventricular tachycardia; atrial fibrillation controlled on medication is not exclusion nor are infrequent or unifocal ectopic beats
* Current QTc prolongation as a result of medication will require discontinuation of that medication; the patient can be reassessed after discontinuation, provided this is medically appropriate, after 2 weeks or five half-lives of the drug have passed whichever is longer
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch blocks (LBBB)
* QTc with Bazett's correction that is unmeasurable, or exceeds 480 msec on screening electrocardiogram (ECG); if a subject has QTc > 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart); the average QTc from the three screening ECGs must be < 480 msec in order for the subject to be eligible for the study
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce cytochrome P450 3A4 (CYP3A4) function
* Hypertension not controlled by medical therapy
* Currently active diarrhea
* Women who are currently pregnant or breast feeding
* Receipt of any investigational agent, chemotherapy or radiation therapy within 21 days prior to Study Day 1
* Any unresolved non-hematologic toxicity greater than CTCAE grade 1 from previous anti-cancer therapy (other than alopecia)
* Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy
* Grade 2 or greater peripheral neuropathy
* Previous or current malignancies within the last 3 years, with the exception of in situ carcinoma of the cervix, adequately treated carcinoma of the skin, small renal masses, and adequately treated localized prostate cancer; other cancers that are highly likely to be cured (cure rate of 75% or greater) may be included at the discretion of the Principal Investigator
* History of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* Patients with brain metastasis can only be included if they were treated more than 4 weeks prior to enrollment; subjects with treated brain metastases must have a post treatment brain magnetic resonance imaging (MRI) showing no further progression of prior lesions AND no new metastatic lesions; subjects will be ineligible if they have any ongoing symptoms from brain metastases or if there continues to be radiographic evidence of cerebral edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06-13 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, M.D., Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 15
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: Defined as the time period from the start of treatment and documented progression or death without documentation of progression. Summarized with Kaplan-Meier curves. The median will be estimated using a non-parametric method.
Time Frame: At 12 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 15
months | 1.4 [1.1 to 2.1]

2. Secondary Outcome: Incidence Grade 3 or Higher Serious Adverse Events (SAE)
Description: Serious Adverse Events will be assessed according to CTCAE version 4.0
Time Frame: Weeks 1, 4, 7, 10, 13, 16, 19, 22 and then every 6 months for up to 2 years
Measure: Number; unit: Events
Arm/Group | Treatment
Number analyzed (Participants) | 15
Events | 22

ADVERSE EVENTS:
Time Frame: 3 years, 3 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 11/15
Serious Adverse Events (participants affected / at risk) | 15/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=15)
Anemia (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Neutrophil count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=15)
Anemia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 10
Fever (General disorders) | 1
Pain (General disorders) | 2
White blood cell decreased (Investigations) | 3
AST/ALT (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2013-05-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT01382706/Prot_000.pdf